CLINICAL TRIAL: NCT00556491
Title: Minocycline to Prevent Acute Kidney Injury After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarek M. El-Achkar (Other)
Collaborators: Satellite Healthcare (Other); Triax Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Tarek M. El-Achkar, Associate Professor, St. Louis University
Organization: St. Louis University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15087
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Kidney Failure, Acute; Acute Kidney Insufficiency
Keywords: renal; kidney; injury; acute; bypass; cardiac; minocycline; prevention; Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury; Wounds and Injuries; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- minocycline (Active Comparator)
  Interventions: Drug: minocycline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: minocycline — given at least for 4 doses (200mg initially then 100mg every 12 hours until surgery)with maximum of 14 doses
  Arms: minocycline
Drug: placebo — placebo will be given for at least 4 doses pre-op to a maximum of 14 doses
  Arms: placebo

SUMMARY:
This study proposes to investigate whether treatment with minocycline pre-operatively in patients with mild to moderate chronic kidney disease undergoing cardiac surgery will reduce the occurence of kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* planned CABG or valvular surgery with cardiopulmonary bypass
* Serum creatinine available (within 30 days)
* Estimated GFR 15-90ml/min using the abbreviated MDRD formula (CKD stages 2-4)

Exclusion Criteria:

* Emergent or urgent surgery (to be performed within the next 36 hours)
* End stage renal disease, or GFR < 15ml/min (CKD stage 5)
* Estimated GFR>90ml/min (CKD stage 1 or no CKD)
* Ongoing infection by positive blood, urine or sputum cultures or pneumonia on CXR
* Allergy to minocycline or tetracyclines
* inability to take oral medications
* use of preoperative vasopressor agents at therapeutic doses
* Pregnant or lactating females
* Advanced liver disease by history or exam(cirrhosis, ascitis, jaundice)
* Rising creatinine meeting the definition of acute kidney injury prior to surgery
* Neurologic signs or symptoms or history of increased intracranial pressure
* current participation in another research study involving an investigational drug or device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M El-Achkar, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Result] Golestaneh L, Lindsey K, Malhotra P, Kargoli F, Farkas E, Barner H, Qazi R, Schmidt A, Rauchman M, Al-Aly Z, Johnson R, Martin K, Dagher P, Friedman A, El-Achkar TM. Acute kidney injury after cardiac surgery: is minocycline protective? J Nephrol. 2015 Apr;28(2):193-9. doi: 10.1007/s40620-014-0152-2. Epub 2014 Oct 28. PMID 25348221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 20 (January 2008) | 20
Completed | 19 | 19
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.9) | 60.8 (11.5) | 62 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
kidney function [Mean (Standard Deviation); unit: ml/min] — Estimated GFR (MDRD)
  ml/min | 71.9 (26.4) | 77.3 (27.4) | 74.3 (26.9)

OUTCOME MEASURES:

1. Primary Outcome: Development of Post-operative Acute Kidney Injury
Description: Participants who develop a Creatinine increase by 0.3 mg/dl (AKIN definition) in any 48 hours time period, within 5 days post-operatively
Time Frame: up to 5 days post cardiac surgery
Measure: Number; unit: participants meeting primary oputcome
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
participants meeting primary oputcome | 10 | 7

2. Secondary Outcome: Post Operative Hospital Days
Time Frame: 30 days post-operative
Measure: Mean (Standard Error); unit: days
Groups:
- Minocycline; Placebo: Post Op hospital days
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
days | 8.7 (3.8) | 9.8 (7.2)

3. Secondary Outcome: On Vent >48 Hours
Description: on ventilator > 48 hours
Time Frame: 30 days post op
Measure: Number; unit: percentage of participant per group
Groups:
- Minocycline; Placebo: On vent > 48 hours
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
percentage of participant per group | 15.8 | 26.3

4. Secondary Outcome: Infections Post Operative
Time Frame: 30 days post operative
Measure: Count of Participants; unit: Participants
Groups:
- Minocycline; Placebo: Infections post-operative
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 2 | 3

5. Secondary Outcome: Stroke Post Operative
Time Frame: 30 days post op
Measure: Count of Participants; unit: Participants
Groups:
- Minocycline: Stroke post-op
- Placebo: stroke post op
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 2 | 0

6. Secondary Outcome: Re-operation
Time Frame: 30 days post-operative
Measure: Count of Participants; unit: Participants
Groups:
- Minocycline; Placebo: re-operation
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Minocycline | Placebo
Serious Adverse Events (participants affected / at risk) | 4/19 | 3/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=19) | Placebo (N=19)
Stroke (Vascular disorders) | 2 | 0
Death (Cardiac disorders) | 0 | 2 — Death within 30 days post-op
Reop (Cardiac disorders) | 2 | 1 — Need for reoperation within 30 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes